CLINICAL TRIAL: NCT00286923
Title: Modulation of the Excitability of the Occipital Cerebral Cortex Using Topiramate
Brief Title: Does Topiramate Adjust the Excitability of the Brain in Migraine Sufferers?
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Emerald City Headache Organization (Other)
Collaborators: Ortho-McNeil Neurologics, Inc. (Industry)
Other Study IDs: CAPSS 347
Record Dates: First submitted 2006-02-02; First posted 2006-02-06 (Estimated); Last update posted 2006-02-14 (Estimated); Status verified 2006-02

CONDITIONS: Migraine; Chronic Headache
Keywords: migraine; chronic headache; hyperexcitability; Magnetic stimulation
MeSH Terms: conditions — Migraine Disorders; Headache Disorders | interventions — Topiramate

INTERVENTIONS:
Drug: Topiramate

SUMMARY:
The purpose of the study is to determine by the use of non-invasive magnetic stimulation if the medication Topiramate adjusts the excitability of the migraine sufferer's brain.

Previous studies have shown the migraine sufferer's brain is more excitable. The magnetic stimulation device has given us a way to look at excitability and to see if it changes at the same time that a headache diary shows if the pattern or severity of headaches changes with the administration of the drug Topiramate.

It is expected that as migraine sufferers have fewer headaches with topiramate the testing with magnetic stimulation will show that their brains are less excitable and that if the topiramate does not change the character of headaches then the pattern of excitabilty would not change from the baseline test before medication is started.

DETAILED DESCRIPTION:
We propose a clinic-based study to test the hypothesis that topiramate modulates the excitability of the occipital cortex in migraine. Subjects between 18 and 55 years old, who have migraine with aura according to IHS criteria will be recruited from the headache clinic. All eligible subjects will have occipital cortex stimulation using the Magstim 200 apparatus. Magnetic brain stimulation will be performed using the 95 mm round coil of the Magstim 200 stimulator. All subjects will be provided ear plugs to prevent possible noise damage to the ear. The recordings will be conducted in a semi-darkened room. Subjects will be asked to focus on the center of a dark screen. A 95 mm diameter circular coil will be applied to the occipital scalp in the midline, 7 cm anterior to the inion. Stimulator intensity will be increased in 10% increments until the subjects report seeing phosphenes (bright scintillating scotomata in the subjects visual field generated by occipital cortical stimulation) or until a maximum of 100% intensity is reached. generated by occipital cortical stimulation) or until a maximum of 100% intensity is reached. Stimulation intensity will be fine tuned to determine the threshold at which phosphenes can be barely seen. In those subjects who do not report seeing phosphenes till 100% intensity, the stimulator will be moved in 1 cm steps to try to define an optimum point for stimulation. No more than 20 stimulations will be given and the frequency shall be kept to less than 5/min. The threshold at which phosphenes are generated will be recorded. To assess inhibitory function of the occipital cortex a visual suppression method will be utilized. Timed TMS impulses usually 10% above phosphene threshold or where suppression is noted will be delivered. Subjects will be asked to report letters projected at a fixed luminance on the screen. Visual suppression will be calculated based on the number of errors the subjects make using an automated analysis. The study procedure will be repeated after the patients have taken topiramate at gradually increasing doses and have achieved stable dose for one month. Patients will be placed on 25 mg at night for 1 week, increased to 25 mg B.I.D. for one week and then maintained at 50 mg B.I.D.

d. There will be no placebo in the study. e. Topiramate will be used in the study.

ELIGIBILITY:
Inclusion Criteria:

Subjects 18 to 55 years old with migraine headaches as defined by the International Headache Society (IHS).

Subjects must be willing to take topiramate for migraine prophylaxis

Exclusion Criteria:

1. Subjects with frequent tension headaches 2. Subjects with ill-defined head pain 3. Unable to be weaned off other headache prophylaxis. 4. Requiring daily use of centrally-acting medications. 5. Pregnant, lactating and women not on adequate birth control measures. 6. Subjects with a personal or family history of seizures of any type. 7. History of head injury or brain surgery. 8. Cardiac pacemakers or any other implanted electronic device. 9. Subjects with history of headaches or with history of tension-type headaches recurring >1/month and relieved by over the counter medications.

-

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10
Dates: Start 2006-02; Study Completion 2006-08

CONTACTS AND LOCATIONS:
Overall Officials: Sheena K. Aurora, M.D., Principal Investigator — Emerald City Headache Organization
Locations (1):
- Swedish Headache Clinic, Seattle, Washington, United States

REFERENCES:
- [Background] Aurora SK, Barrodale P, Chronicle EP, Mulleners WM. Cortical inhibition is reduced in chronic and episodic migraine and demonstrates a spectrum of illness. Headache. 2005 May;45(5):546-52. doi: 10.1111/j.1526-4610.2005.05108.x. PMID 15953273
- [Background] Aurora SK, Cao Y, Bowyer SM, Welch KM. The occipital cortex is hyperexcitable in migraine: experimental evidence. Headache. 1999 Jul-Aug;39(7):469-76. doi: 10.1046/j.1526-4610.1999.3907469.x. PMID 11279929
- [Background] Aurora SK, Ahmad BK, Welch KM, Bhardhwaj P, Ramadan NM. Transcranial magnetic stimulation confirms hyperexcitability of occipital cortex in migraine. Neurology. 1998 Apr;50(4):1111-4. doi: 10.1212/wnl.50.4.1111. PMID 9566403